CLINICAL TRIAL: NCT04464603
Title: Impact of a Shared Decision-making mHealth Tool on Caregivers' Team Situational Awareness, Communication Effectiveness, and Performance During Pediatric Cardiopulmonary Resuscitation: a Randomized Controlled Trial
Brief Title: Impact of a mHealth Supportive Tool on Cardiopulmonary Resuscitation' Situational Awareness
Acronym: InterFACE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pediatric Clinical Research Platform (Other)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Johan Siebert, MD, MD, Deputy Head, Pediatric Clinical Research Platform
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: InterFACE
Record Dates: First submitted 2020-07-02; First posted 2020-07-09 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Cardiopulmonary Arrest; Pediatric ALL; Resuscitation
Keywords: Information technologies; Situation Awareness; Teamwork; Leadership; Mobile applications; Biomedical Technology
MeSH Terms: conditions — Heart Arrest; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: A prospective, single center, randomized controlled trial
Who Masked: Participant
Masking Description: Blinding to the outcomes will be maintained during recruitment to minimize preparation bias. Allocation concealment will be ensured with an allocation software and will not be released until the participants start the scenario. A post-scenario video review will be done without blinding by two reviewers, but undertaken independently with each blinded to the other's reviews. In the case of disagreement, a third independent evaluator will help reach a consensus. The data analyst will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (InterFACE) (Experimental): Participants that will use the mHeath InterFACE tool during the simulation-based pediatric scenario.
  Each participant will have to do 2 consecutive scenarios (PALS, ATLS).
  Interventions: Device: InterFACE (mHealth tool)
- Arm B (Conventional methods) (Active Comparator): Participants that will use conventional methods during the simulation-based pediatric scenario.
  Each participant will have to do 2 consecutive scenarios (PALS, ATLS).
  Interventions: Other: Conventional methods

INTERVENTIONS:
Device: InterFACE (mHealth tool) — Participants will be asked to perform consecutively two 20-min highly realistic, scripted CPR scenarios (first: PALS-based scenario, second: ATLS-based scenario) on a high-fidelity WiFi manikin.
  Within each scenario, 3 separate "freeze" periods will occur at random points in time to assess the shared and complementary Situation Awareness of each team member individually regarding the CPR in progress at that exact moment in time. The scenarios will be standardized to strictly follow the 2018 AHA algorithms and the 2018 ATLS guidelines.
  Both scenarios will be completed in the same order and the procedure will be standardized across all teams to follow the same chronological progression and range of difficulty in order to ensure that each participant is exposed to exactly the same case, with similar challenges in technical and non-technical skills.
  Participants allocated to Arm A will not be allowed to use any other cognitive support.
  Arms: Arm A (InterFACE)
Other: Conventional methods — Participants will be asked to perform consecutively two 20-min scripted CPR scenarios (PALS and ATLS-based scenario) on a high-fidelity WiFi manikin.
  Within each scenario, 3 separate "freeze" periods will occur at random points in time to assess the shared and complementary Situation Awareness of each team member individually regarding the CPR in progress at that exact moment in time. The scenarios will be standardized to strictly follow the 2018 AHA algorithms and 2018 ATLS guidelines.
  Both scenarios will be completed in the same order and the procedure will be standardized across all teams to follow the same chronological progression and range of difficulty in order to ensure that each participant is exposed to exactly the same case, with similar challenges in technical and non-technical skills.
  Participants allocated to group B will be allowed to use the PALS pocket reference cards and a conventional calculator, but not any other cognitive support or mHealth tool.
  Arms: Arm B (Conventional methods)

SUMMARY:
This study will be a prospective, single-center, randomized controlled trial in a tertiary pediatric emergency department with two parallel groups of voluntary pediatric physicians and nurses. The impact of a mHealth supportive tool will be compared with conventional communication methods on situational awareness, leadership, team communication effectiveness and performance during standardized, simulation-based, pediatric in-hospital cardiac arrest scenario using a high-fidelity manikin. Thirty-six participants will be randomized (1:1). The primary endpoint is the situational awareness score measured with the situation awareness global assessment technique (SAGAT) instrument.

DETAILED DESCRIPTION:
Effective team communication, coordination, and situational awareness by cardiac arrest team members are critical components to deliver optimal cardiopulmonary arrest resuscitation care. But the complexity of care during cardiopulmonary resuscitation (CPR), numerous providers involved, miscommunication, and exogenous factors can all contribute to wresting patients care, thus jeopardizing their survival. The aim of this trial is to investigate whether a mHealth supportive tool (the interconnected and focused mobile apps on patient care environment [InterFACE]) developed as a collaborative platform to support CPR providers in real-time and share patient-centered information would increase situational awareness during pediatric CPR and improve team communication and performance.

This clinical trial will be a prospective, single-center, randomized controlled trial in a tertiary pediatric emergency department (>33,000 consultations/year) with two parallel groups of voluntary pediatric emergency fellows, residents and nurses.

Situational Awareness (SA), leadership, communication skills and team performance will be compared using a shared mHealth supportive tool ("InterFACE", group A) or conventional team interactions (group B) during standardized simulation-based pediatric in-hospital cardiac arrest scenario (p-IHCA) and life-threatening trauma scenarios using a high-fidelity manikin. InterFACE consists of a dual, interconnected mHealth tool composed primarily of a mobile device app, namely "Guiding Pad" (PMID: 32292179), interfaced to a remote large liquid crystal display (LCD) screen installed in the shock room and situated above the patient's head.

Thirty-six participants will be randomized 1:1 (each team will comprise six participants, i.e. a total of 6 teams). The teams will be asked to perform consecutively two 20-min highly realistic, scripted CPR scenarios on a high-fidelity WiFi manikin (Laerdal SimBaby, Laerdal Medical, Stavanger, Norway) using either the mHealth tool or conventional methods. The scenarios will be standardized to strictly follow the 2018 AHA algorithms and the 2018 ATLS guidelines.

In this simulation-based study, each team member will answer the SAGAT queries specific to their roles. Leadership will be measured with the resuscitation team leader evaluation (RTLE) instrument. Effective teamwork and communication will be measured with the team emergency assessment measure (TEAM) instrument. The SUS instruments will be used to measure the usability of the mHealth tool. For the trauma scenario, the modified non-technical skills scale for trauma (T-NOTECHS) will not be used due to the serious risk of assessment bias with this instrument, as emphasized by the consensus-based standards for the selection of health measurement instruments (COSMIN).

Data collection will be carried out by the responsive simulator detectors (Laerdal SimBaby) and the two GoPro video cameras. The set-up of both cameras will be standardized. The recorded videos will be safely stored in duplicate on secured hard-disk drives in a locked room. As all scenarios will be fully video-recorded, all actions, communications and interactions will be recorded and later scored by two raters to allow outcomes analysis and for the calculation of interrater reliability. All actions performed with the app will be automatically saved locally in log files for further analysis. This study offers the major advantage to observe a unique 60-min period per resuscitation team. Therefore, neither follow-up nor retention plans will be necessary. The resuscitation algorithm is highly standardized and deviation from the algorithm is a parameter of interest in this study. Data collection will be carried out using the REDCap database (REDCap, Vanderbilt University, Nashville, TN, USA).

This clinical trial will assess the impact of a collaborative mHealth tool to increase situational awareness and effective team communication during in-hospital pediatric resuscitation. As research in this area is scarce, the results generated from this study will be of great importance and may be sufficient to change and improve in-hospital pediatric emergency care practice in an era of communication technologies.

ELIGIBILITY:
Inclusion Criteria:

* Any physician performing a fellowship in the pediatric emergency department.
* Any postgraduate residents pursuing a <5 years residency in pediatrics.
* To be registered nurses from the PED.
* To have previously completed a standardized 15-min introductory course on the use of the InterFACE tool dispensed by the study investigators.
* Participation agreement

Exclusion Criteria:

* To have not undergone the standardized 15-min introductory course on the use of the InterFACE tool dispensed by the study investigators.
* Participation to a simulation in the past month is an exclusion criterion to avoid a recent training effect.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Situational awareness | 40 minutes
  Situational awareness (SA) will be measured using retrospective video review by the SA global assessment technique (SAGAT) instrument for each scenario, both as the score of each SAGAT at an individual level and at the team level (given as the sum of individual SAGAT scores for each team; TSAGAT). The SAGAT responses for categorical variables will be scored as either correct (1) or incorrect (0) by two of the investigators, irrespective of whether they agreed completely with the true answer. For numerical responses, answers will be considered correct based upon a 10% pre-defined tolerance range settled by the research investigators around the true value. The scores will be expressed as percentages in conjunction with absolute n/N values. Higher SA scores will denote higher SA.

SECONDARY OUTCOMES:
Resuscitation team leader evaluation | 40 minutes
  Leadership will be measured using the 12-item RTLE instrument developed by Grant et al. that encompasses four leadership concepts: (1) the physical and verbal leader's position; (2) communication and delegating skills; (3) ability to assess, adapt and anticipate; and (4) ability to ask for internal and external help. This instrument comprises 12 items rated on a 4-point Likert scale from 0 (not performed) to 3 (performed well) to score leadership and communication skills. A not applicable (N/A) category is also available for those items not relevant to the scenario. For the purpose of this trial, items 1 and 12 will be removed as the leader will be clearly identified from the beginning of the scenario and teams will not be advised to ask for external help. Therefore, the total item score will range from 0 to 30.
Team Emergency Assessment Measure | 40 minutes
  Teamwork performance will be measured using the 11-item Team Emergency Assessment Measure (TEAM) tool that stands out as the most valid and reliable instrument to use in emergency departments. TEAM comprises 11 items rated on a 5-point Likert scale from 0 (never/hardly) to 4 (always/nearly always), which are summed up into a total item score ranging from 0 to 44. The final score obtained allows to assess the performance of the emergency medical team based on three categories: leadership (items 1 and 2); teamwork (items 3 to 9); and task management (items 10 and 11). Items 8 and 9 relate to SA perception and projection, respectively. Furthermore, the team's overall performance is rated through a twelfth item on a global rating scale of 1 to 10 (higher score denotes better performance).
Medication dosage errors | 40 minutes
  Errors in drug dose administration (in milligrams) will be measured in each allocation group as a deviation from the 2018 AHA PALS cardiac arrest algorithm. An emergency medication dose administration error is defined as a deviation from the correct weight dose of more than 10%. Errors will be also measured both as the percentage deviation from the amount of delivered drug compared with the correct weight dose as prescribed by the physician and the absolute deviations from that dose.
  Moreover, defibrillations (in Joules) and the number of shocks will be also measured during the first scenario. For the second scenario, errors in fluid resuscitation volumes (in milliliters) will be measured as a deviation from the 2018 ATLS guidelines.
Time to critical life-saving maneuvers | 40 minutes
  The elapsed time in seconds between the end of the clinical statement by the study investigator to: (1) cardiac arrest or hypotensive shock recognition; (2) initiation of chest compression; (3) time to each defibrillation attempt; (4) time to administration of intravenous drugs, volume expansion with 0.9% sodium chloride or blood transfusion; and (5) time interval between defibrillation attempts will be measured.
System usability scale | 10 minutes
  Usability testing of the mHealth tool InterFACE will be assessed using the System Usability Scale (SUS) instrument. The SUS instrument consists of a 10-item questionnaire with five response options for each item, based on their level of agreement ranging from 1 (strongly disagree) to 5 (strongly agree). For odd-numbered statements 1, 3, 5, 7, 9 (positively-worded items), the score contribution is equal to the scale position minus 1. For even-numbered statements 2, 4, 6, 8, 10 (negatively-worded items), the score contribution is equal to 5 minus the scale position. Each score contribution will fall within the range of 0 to 4. The participant's scores for each item are then added up together and multiplied by 2.5 to convert the original scores of 0-40 to 0-100.
Team effectiveness | 40 minutes
  Team effectiveness will be also measured as the time spent by the team to achieve the pre-designed goals set out by the AHA for the PALS course and the American College of Surgeons for the ATLS course.
Stress perceived and satisfaction | 10 minutes
  A 3-item questionnaire using a 10-point Likert scale will be provided to the participants to measure their perceived stress and satisfaction about the preparation method used during the resuscitation scenario.
  The questionnaire measures (1) the stress perceived before the scenario starts (On a scale from 1 to 10, how stressed are you now?), (2) the overall stress perceived at the end of the scenario (On a scale of 1 to 10, how stressed [maximum reached] were you during the scenario?), and (3) the satisfaction about the supportive method used during the resuscitation scenario (On a scale of 1 to 10, how satisfied were you with your supported experience?)
  Scale ranges: from 0 (minimum score) to 10 (maximum score), increments are integers between 0 to 10. For stress, higher values represent a worse score, whereas for satisfaction higher values represent a better score. No subscales will be combined.

CONTACTS AND LOCATIONS:
Overall Officials: Johan N Siebert, MD, Principal Investigator — Geneva Children's Hospital, Geneva University Hospitals, Geneva, Switzerland
Locations (1):
- Geneva Children's Hospital, Geneva University Hospitals, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
IPD will be deidentified and the study investigators will house the data locally on secure hard disk drives at the Geneva Children's Hospital. The datasets used or analyzed during the current trial will be available from the corresponding author upon reasonable request. Only deidentified/anonymized data will be shared.
Supporting Information: Study Protocol
Time Frame: Available from 1 month to 10 years after trial publication.
Access Criteria: From the corresponding author upon reasonable request.

REFERENCES:
- [Background] Siebert JN, Lacroix L, Cantais A, Manzano S, Ehrler F. The Impact of a Tablet App on Adherence to American Heart Association Guidelines During Simulated Pediatric Cardiopulmonary Resuscitation: Randomized Controlled Trial. J Med Internet Res. 2020 May 27;22(5):e17792. doi: 10.2196/17792. PMID 32292179
- [Derived] Ehrler F, Sahyoun C, Manzano S, Sanchez O, Gervaix A, Lovis C, Courvoisier DS, Lacroix L, Siebert JN. Impact of a shared decision-making mHealth tool on caregivers' team situational awareness, communication effectiveness, and performance during pediatric cardiopulmonary resuscitation: study protocol of a cluster randomized controlled trial. Trials. 2021 Apr 13;22(1):277. doi: 10.1186/s13063-021-05170-3. PMID 33849611